CLINICAL TRIAL: NCT02570542
Title: A Multi-center Randomized Phase II Study of the Impact of CD34+ Cell Dose on Absolute Lymphocyte Count Following High-Dose Therapy and Autologous Stem Cell Transplantation for Relapsed and Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Study of the Impact of CD34+ Cell Dose on Absolute Lymphocyte Count Following High-Dose Therapy and Autologous Stem Cell Transplantation for Relapsed and Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Columbia University (Other); Endeavor Health (Other); University of Rochester (Other); Medical College of Wisconsin (Other); University of Nebraska (Other); Sanofi (Industry); University Hospitals Seidman Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-193
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL); Relapsed Diffuse Large B-cell Lymphoma (DLBCL); Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Keywords: CD34+ Cell Dose; Autologous Stem Cell Transplantation; 15-193
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Leukapheresis; plerixafor; Carmustine; Etoposide; Cytarabine; Melphalan

ARMS (2):
- 3-4 x 10^6 CD34+ stem cells/kg (Active Comparator): Patients will receive standard supportive measures (including: growth factor support post-HDT/ASCT, antimicrobial prophylaxis, red blood cell and platelet transfusion and treatment for neutropenic fever) as per institutional guideline practices.
  Interventions: Procedure: leukapheresis; Drug: Plerixafor; Drug: carmustine, etoposide, cytarabine, melphalan; Procedure: Autologous Stem Cell Transplantation
- 6-8 x10^6 CD34+ stem cells/kg (Experimental): Patients will receive standard supportive measures (including: growth factor support post-HDT/ASCT, antimicrobial prophylaxis, red blood cell and platelet transfusion and treatment for neutropenic fever) as per institutional guideline practices.
  Interventions: Procedure: leukapheresis; Drug: Plerixafor; Drug: carmustine, etoposide, cytarabine, melphalan; Procedure: Autologous Stem Cell Transplantation

INTERVENTIONS:
Procedure: leukapheresis
Drug: Plerixafor — Following enrollment, patients will be CD34+ stem cell mobilized at the discretion of the treating attending physician with the plerixafor for a maximum of 4 apheresis days, for the achievement of ≥ 7 x106 CD34+ cells/kg.
Drug: carmustine, etoposide, cytarabine, melphalan — Carmustine 300 mg/m2 day -6 Etoposide 100 mg/m2 q12hrs x 8 doses day - 5 thru day -2 Cytarabine 100 mg/m2 q12hrs x 8 doses day - 5 thru day -2 Melphalan 140 mg/m2 day -1 BEAM dosages may be adjusted per institutional dose adjustments based on body weight.
  Other Names: BEAM chemotherapy
Procedure: Autologous Stem Cell Transplantation

SUMMARY:
The purpose of this study is to study the impact of stem cell dose on outcome after autologous transplant.

DETAILED DESCRIPTION:
Following enrollment, patients will be CD34+ stem cell mobilized at the discretion of the treating attending physician with the plerixafor for the achievement of >6 x10^6 CD34+ cells/kg. The patients that fail to mobilize >6 x10^6 CD34+ cells/kg will not be randomized and will subsequently be followed for disease progression and overall survival.. Patients with >6 x10^6 CD34+ cells/kg cryopreserved on study will be admitted to the hospital for planned ASCT. Patients will be randomly infused with either 3-4 x 10^6 CD34+ stem cells/kg or 6-8 x10^6 CD34+ stem cells/kg on d0 per study randomization. The cell dose ranges within the two groups allows variability within aliquots of cells at the time of cryopreservation. Patients will receive standard supportive measures (including: growth factor support post-HDT/ASCT, antimicrobial prophylaxis, red blood cell and platelet transfusion and treatment for neutropenic fever) as per institutional guideline practices.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosed with relapsed or refractory de novo DLBCL or follicular lymphoma transformed to DLBCL to one previous line of anthracycline-containing chemotherapy
* KPS ≥ 70
* Complete or partial response by IWG Working Group or ICML Criteria to maximum of one salvage line of chemotherapy without pre-HDT/ASCT salvage radiotherapy.
* Eligible for high-dose therapy and autologous stem-cell rescue

  * Serum creatinine ≤ 1.5 mg/dL, or if creatinine >1.5 mg/dL, calculated creatinine clearance of ≥50 mL/min by 24 hour creatinine clearance or CKD-EPI.
  * Last cycle of most recent salvage therapy within 8 weeks of enrollment
* Total bilirubin < 2.0 mg/dL

  o If Gilbert"s disease is suspected and total bilirubin > 2.0 mg/dL, direct bilirubin must be < 2.0 mg/dL
* Females of childbearing potential and males must agree to use an acceptable form of contraception per institutional practices.

Exclusion Criteria:

* Disease progression by IWG Working Group or ICML Criteria since last therapy
* Prior autologous or allogeneic stem cell transplantation
* HIV infection
* Comorbid condition(s) which, in the opinion of the attending physician and/or MSKCC Principal Investigator, will preclude stem cell mobilization and/or high-dose therapy with autologous stem cell rescue
* Treatment plan that includes post-transplant maintenance therapy
* Salvage therapy that includes involved field radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | at +/- 2 weeks
  equals date of progression/death - date of Autologous Stem Cell Transplantation

SECONDARY OUTCOMES:
the impact of CD34+ cell dose on lymphocyte subset recovery | day 15
  (ALC15) post HDT-ASCT Accordingly, each subject will be classified as a responder (i.e., recovery) or non-responder.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (14):
- United States (14):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge (Consent and Follow-Up Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow up Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow Up Only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow-up Only), Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health (Data collection only), Manhasset, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow up Only), Uniondale, New York
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Transplant Institute, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/